CLINICAL TRIAL: NCT00201838
Title: A Phase I/II Study of Etanercept and Gemcitabine in Patients With Advanced Stage and Chemotherapy Naive Pancreatic Adenocarcinoma
Brief Title: Etanercept and Gemcitabine in Patients With Advanced, Chemotherapy Naive Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0041
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Pancreatic Neoplasms; Adenocarcinoma
Keywords: Advanced Stage; Chemotherapy Naive
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Gemcitabine; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients received entanercept 25 mg subcutaneously twice weekly with gemcitabine.
  Interventions: Drug: Gemcitabine; Drug: Etanercept
- Arm II (Active Comparator): Patients with pancreatic cancer for which treatment with gemcitabine as a single agent is planned will be asked to participate in this trial as a control group.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — The starting dose will be 1000mg/m2 IV, weekly x 7 with a one week rest followed by weekly x 3 with one week rest for the remainder of treatment.
  Other Names: Gemzar®
Drug: Etanercept — Etanercept will be self administered subcutaneously by patients with injections 11 prepared by the investigational pharmacy, beginning 7 days prior to the first dose of gemcitabine and continued twice weekly for the duration of the study.
  Other Names: Enbrel
  Arms: Arm I

SUMMARY:
The aims of this protocol are:

1. To study the safety and tolerability of the combination of etanercept and gemcitabine in patients with advanced pancreatic cancer:
2. To estimate the anti-tumor effect as measured by the proportion of patients free of disease-progression at six months after treatment initiation.

DETAILED DESCRIPTION:
Rationale: The standard treatment for pancreatic cancer is gemcitabine. This study combines gemcitabine with etanercept, a drug that binds with tumor necrosis factor (TNF) molecules and blocks their activity through inhibiting their interaction with cell surface TNF receptors. TNF is the name for a protein in the body that often helps fight foreign substances. However, research suggests that pancreatic tumors develop resistance to TNF and then use it to support cancer growth. Combining etanercept, a TNF inhibitor, with gemcitabine is a novel approach to advanced pancreatic cancer. Because etanercept has not been tested in combination with gemcitabine, a Phase I study will be conducted first to identify the safest dosage of etanercept, and then a Phase II study will evaluate the efficacy of this combination.

Purpose: This study is evaluating the safety of etanercept and gemcitabine for advanced pancreatic cancer in Phase I, and the efficacy of etanercept and gemcitabine for this condition in Phase II. TNF and other inflammatory markers will also be measured in the study.

Treatment: Patients in this study will receive gemcitabine and etanercept. Gemcitabine will be administered through an intravenous infusion weekly for seven weeks followed by one week of rest. Additional treatments with gemcitabine will be given for three weeks followed by one week of rest. Patients will administer etanercept to themselves through a small injection underneath the skin twice each week. Six patients will initially be enrolled in Phase I. If severe side effects appear in at least two patients in Phase I, then additional patients will be enrolled and treated with lower dosages of gemcitabine. When the treatments do not produce unacceptable side effects, the Phase I portion of the study will end and Phase II will begin enrolling patients. Patients in the Phase II portion of the study will also receive gemcitabine and etanercept at the safest dosages identified in Phase I. Several tests and exams will be given throughout both portions of the study to closely monitor patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have pathological diagnosis recurring or metastatic Pancreatic Adenocarcinoma
* No prior chemotherapy, immunology treatments or hormonal treatments
* Measurable disease
* Must be >18 years old
* ONLY CONTROL ARM IS OPEN TO ACCRUAL

Inclusion Criteria:

* Pregnant and nursing mothers.
* Psychiatric disorders that would interfere with consent ability.
* Patients with known brain or leptomeningeal disease.
* Patients with history of myocardial infarction with in six previous months.
* Any concurrent illness that would constitute a hazard to participation in study.
* Known sensitivity to gemcitabine or etanercept.
* Prior treatment with etanercept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2001-07; Primary Completion 2006-10 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villalona, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Wu C, Fernandez SA, Criswell T, Chidiac TA, Guttridge D, Villalona-Calero M, Bekaii-Saab TS. Disrupting cytokine signaling in pancreatic cancer: a phase I/II study of etanercept in combination with gemcitabine in patients with advanced disease. Pancreas. 2013 Jul;42(5):813-8. doi: 10.1097/MPA.0b013e318279b87f. PMID 23429495
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: combination of gemcitabine and etanercept
  Gemcitabine: The starting dose will be 1000mg/m2 IV, weekly x 7 with a one week rest followed by weekly x 3 with one week rest for the remainder of treatment.
  Etanercept: Etanercept will be self administered subcutaneously by patients with injections 11 prepared by the investigational pharmacy, beginning 7 days prior to the first dose of gemcitabine and continued twice weekly for the duration of the study.
- Control Group: Patients received gemcitabine alone
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 30 | 8
Treatment Cohort | 30 | 8
Completed | 30 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Interventional Arm: Patients received Etanercept with gemcitabine
- Control Arm: Patients received Gemcitabine alone
- Total: Total of all reporting groups
Arm/Group | Interventional Arm | Control Arm | Total
Number analyzed (Participants) | 30 | 8 | 38
Age, Continuous [Median (Full Range); unit: years] | 59 [46 to 81] | 59 [46 to 75] | 59 [46 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 16 | 3 | 19
Region of Enrollment [Number; unit: participants]
  United States | 30 | 8 | 38
Metastatic Site [Number; unit: patients]
  Liver only | 16 | 0 | 16
  Liver + other | 10 | 6 | 16
  other site | 4 | 2 | 6
ECOG Performance Status (PS) [Number; unit: patients] — Eastern Cooperative Oncology Group (ECOG)
  patients
    PS 0 (Fully active) | 7 | 3 | 10
    PS 1 (Restricted in physical activity) | 21 | 5 | 26
    PS 2 (Ambulatory and capable of selfcare) | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumor Effect as Measured by the Proportion of Patients Free of Disease-progression at Six Months After Treatment Initiation
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Percentages were calculated by a Kaplan Meier analysis.
Time Frame: up to 6 months
Population: 5 patients of the experimental group were non evaluable and 2 patients in the control group were non evaluable for disease progression.
Measure: Number; unit: percent of patients with PFS
Groups:
- Experimental Group: Patients received etanercept 25mg subcutaneously twice-weekly with gemcitabine
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 25 | 6
percent of patients with PFS | 28 | 14

2. Secondary Outcome: Number of Patients With Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: up to 12 months
Population: 2 patients in the control group were non evaluable for disease response due to patient withdrawal and another no baseline imaging for comparison.
  5 patients in experimental group were non evaluable for response.
Measure: Number; unit: percentage of patients
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 25 | 6
percentage of patients
  Partial Response | 12 | 17
  Stable Disease | 32 | 50

3. Secondary Outcome: Percentage of Patients With Clinical Benefit Response
Description: A clinical benefit was defined by the improvement of at least one parameter over at least 4 weeks, without worsening of any other parameter (change in weight, ECOG performance status, Quality of life).
Time Frame: Up to 12 months
Population: All evaluable patients
Measure: Number; unit: percentage of patients
Groups:
- Experimental Group: Etanercept with gemcitabine
- Control Group: Gemcitabine alone
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 15 | 2
percentage of patients | 33 | 0

4. Secondary Outcome: Median Overall Survival Rates for Patients
Description: Median survival is defined as the time of initiation of the first dose of intervention to the date of death
Time Frame: up to 1 year
Population: all evaluable patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 29 | 8
months | 5.43 [3.30 to 10.23] | 8.1 [3.1 to 20.4]

5. Secondary Outcome: Serial Levels of TNF (Tumor Necrosis Factor) and Other Inflammatory Cytokines
Time Frame: up to 6 months
Population: Compare CBR with responders and non responders with available blood samples.
Measure: Mean (Standard Deviation); unit: delta Ct values
Groups:
- Responders: combination of gemcitabine and etanercept
  Gemcitabine: The starting dose will be 1000mg/m2 IV, weekly x 7 with a one week rest followed by weekly x 3 with one week rest for the remainder of treatment.
  Etanercept: Etanercept will be self administered subcutaneously by patients with injections 11 prepared by the investigational pharmacy, beginning 7 days prior to the first dose of gemcitabine and continued twice weekly for the duration of the study.
- Non Responders: Gemcitabine: The starting dose will be 1000mg/m2 IV, weekly x 7 with a one week rest followed by weekly x 3 with one week rest for the remainder of treatment.
  Etanercept: Etanercept will be self administered subcutaneously by patients with injections 11 prepared by the investigational pharmacy, beginning 7 days prior to the first dose of gemcitabine and continued twice weekly for the duration of the study.
Arm/Group | Responders | Non Responders
Number analyzed (Participants) | 6 | 7
delta Ct values
  IL-10 | 28.04 (1.93) | 26.85 (1.38)
  IL-1b | 16.2 (7.29) | 13.07 (7.44)
  NFkB | 6.03 (4.62) | 4.38 (3.13)
  IL-12 | 35.66 (1.86) | 36.11 (1.24)
  TNF | 26.66 (3.84) | 27.26 (4.82)
  IFN | 28.7 (2.13) | 28.63 (1.55)
  IL-6 | 29.25 (1.31) | 29.29 (1.39)

ADVERSE EVENTS:
Description: Toxicities were graded according to the NCI Common Toxicity Criteria version 3.0. One patient was not evaluable for toxicity in the Experimental Group.
Groups:
- Experimental Group: Patients in the experimental group received etancercept 25 mg subcutaneously twice-weekly with gemcitabine.
- Control Group: Patients in the control cohort received gemcitabine alone.
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/8
Other Adverse Events (participants affected / at risk) | 29/29 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group (N=29) | Control Group (N=8)
Anemia (Blood and lymphatic system disorders) | 20 (20) | 7 (7)
Leukopenia (Investigations) | 12 (12) | 6 (6)
Neutropenia (Investigations) | 9 (9) | 3 (3)
Thrombocytopenia (Injury, poisoning and procedural complications) | 8 (8) | 5 (5)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 14 (14) | 5 (5)
Nausea (Gastrointestinal disorders) | 14 (14) | 6 (6)
Dysgeusia (Nervous system disorders) | 12 (12) | 2 (2)
Constipation (Gastrointestinal disorders) | 9 (9) | 4 (4)
Vomiting (Gastrointestinal disorders) | 8 (8) | 4 (4)
Transaminases (Investigations) | 8 (8) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Edema (Vascular disorders) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Injection reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The interpretation of the results for this study is limited by the relatively small patient sample and correlative samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes